CLINICAL TRIAL: NCT02952261
Title: Three-Dimensional Printing of Navigational Template in Localization of Small Pulmonary Nodule: A Prospective, Randomized, Controlled, Non-inferiority Trial
Brief Title: Application of 3D Printing Technique in Small Pulmonary Nodule Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Chen (Other)
Responsible Party: Sponsor-Investigator, Chang Chen, Chief of thoracic surgery, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k16-284
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Lung Neoplasm; Thoracic Surgery, Video-Assisted
Keywords: Printing, Three-dimensional
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-guided localization (Other): This group of participants received conventional CT-guided lung nodule localization.
  Interventions: Other: CT-guided localization
- template-guided localization (Experimental): Three-dimensional printed template was customized based on participant's computed tomography information. Participants received template-guided lung nodule localization.
  Interventions: Device: template-guided localization

INTERVENTIONS:
Device: template-guided localization — Based on CT data, digital model of the navigational template was created using CAD software and imported to 3D printer. The navigational template serves as a guider to the localizer in lung nodule localization.
  Arms: template-guided localization
Other: CT-guided localization — Percutaneous lung nodule localization was conducted under the real-time guidance of CT scan. This is the conventional method of transthoracic lung nodule localization.
  Arms: CT-guided localization

SUMMARY:
The trial is to evaluate the efficacy and safety of three-dimensional printed navigational template in the clinical application of small peripheral lung nodule localization.

DETAILED DESCRIPTION:
Localization of small lung nodule is challenging due to the difficulty of nodule recognition during VATS. A three-dimensional printed navigational template was designed to aid percutaneous lung nodule localization, and its feasibility has been confirmed in previous study. The trial was conducted to confirm the non-inferiority of template-guided method to conventional CT-guided method in terms of localization accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 19 to 80 years
2. lesions located in peripheral lung tissue which can be removed by wedge resection
3. The maximum diameter of the lesion is no more than 20 mm.
4. Research assistant consulted with the patient's surgeon to confirm the necessity of lung nodule localization
5. Informed consent was signed voluntarily.

Exclusion Criteria:

1. nodule located in the scapula region.
2. there were two or more lung nodules needed to be localized.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, MD,Ph.D, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang L, Li M, Li Z, Kedeer X, Wang L, Fan Z, Chen C. Three-dimensional printing of navigational template in localization of pulmonary nodule: A pilot study. J Thorac Cardiovasc Surg. 2017 Dec;154(6):2113-2119.e7. doi: 10.1016/j.jtcvs.2017.08.065. Epub 2017 Sep 1. PMID 29017792
- [Derived] Zhang L, Wang L, Kadeer X, Zeyao L, Sun X, Sun W, She Y, Xie D, Li M, Zou L, Rocco G, Yang P, Chen C, Liu CC, Petersen RH, Ng CSH, Parrish S, Zhang YS, Giordano R, di Tommaso L; AME Thoracic Surgery Collaborative Group. Accuracy of a 3-Dimensionally Printed Navigational Template for Localizing Small Pulmonary Nodules: A Noninferiority Randomized Clinical Trial. JAMA Surg. 2019 Apr 1;154(4):295-303. doi: 10.1001/jamasurg.2018.4872. PMID 30586136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process was from October 15, 2016 to October 26, 2017. And, the first participant was recruited on October 24, 2016. Until reaching to 40% of prespecified sample size (Janunary 1, 2017) , interim analysis was conducted.
Period: Overall Study
Arm/Group | CT-guided Localization | Template-guided Localization
Started | 100 | 100
Completed | 95 | 95
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-guided Localization | Template-guided Localization | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11) | 54 (15) | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 74 | 147
  Male | 27 | 26 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Smoking history [Count of Participants; unit: Participants]
  YES | 28 | 30 | 58
  NO | 72 | 70 | 142
BMI(body mass index) [Mean (Standard Deviation); unit: Kg/m^2] | 22.9 (2.9) | 22.8 (2.8) | 22.9 (2.8)
FEV1（of percentage predicted） [Mean (Standard Deviation); unit: Percentage predicted FEV1] | 93.6 (13.0) | 94.3 (14.6) | 94.0 (13.8)
Nodule size [Mean (Standard Deviation); unit: mm] — nodule size measured by long-axis diameter
  mm | 9.2 (2.7) | 10.1 (3.0) | 9.7 (2.9)
Nodule location [Count of Participants; unit: Participants]
  right upper lobe(RUL) | 26 | 38 | 64
  right middle lobe(RML) | 9 | 5 | 14
  right lower lobe(RLL) | 26 | 17 | 43
  left upper lobe(LUL) | 22 | 25 | 47
  left lower lobe(LLL) | 17 | 15 | 32
Nodule type [Count of Participants; unit: Participants]
  pure ground glass opacity(GGO) | 55 | 41 | 96
  Mixed ground glass opacity(GGO) | 35 | 50 | 85
  Solid | 10 | 9 | 19
Distance from pleura [Median (Full Range); unit: mm] | 6.5 [0 to 35.9] | 8.5 [0 to 43.9] | 7.8 [0 to 43.9]

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Lung Nodule Localization
Description: Localization accuracy was defined by the localizer deviation between the hookwire and the center of the target nodule. (The deviation was measured using CAD software after downloading the CT images from the Picture Archiving and Communication Systems.)
Time Frame: From the time of completing final CT scan, assessed up to 2 days.
Population: Modified Intention-to-treat analysis (patients who did not receive lung nodule localization were excluded.(n=10))
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CT-guided Localization | Template-guided Localization
Number analyzed (Participants) | 95 | 95
mm | 9.6 (5.8) | 8.7 (6.9)

2. Secondary Outcome: Procedural Duration of the Nodule Localization
Description: Procedural duration was derived from CT scan parameters, which was calculated as the time length between the initial and final scan.
Time Frame: From the time of completing final CT scan, assessed up to 1 hour.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | CT-guided Localization | Template-guided Localization
Number analyzed (Participants) | 95 | 95
min | 9.5 (3.6) | 7.4 (3.2)

3. Secondary Outcome: Radiation Dose
Description: Radiation dosage was read on the monitor screen of CT scanner and converted to effective dosage.
Time Frame: From the time of completing final CT scan, assessed up to 1 hour.
Measure: Mean (Standard Deviation); unit: mGy*cm
Arm/Group | CT-guided Localization | Template-guided Localization
Number analyzed (Participants) | 95 | 95
mGy*cm | 313 (84) | 229 (65)

4. Secondary Outcome: Complication Rate
Description: Pnuemothorax related to lung nodule localization
Time Frame: From the time of completing final CT scan, assessed up to 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-guided Localization | Template-guided Localization
Number analyzed (Participants) | 95 | 95
Participants | 17 | 10

ADVERSE EVENTS:
Time Frame: Adverse event were assessed immediately after lung nodule localization through CT scanning, assessed up to 2 days.
Arm/Group | CT-guided Localization | Template-guided Localization
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/95
Other Adverse Events (participants affected / at risk) | 28/95 | 16/95
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-guided Localization (N=95) | Template-guided Localization (N=95)
pnueumothorax (Surgical and medical procedures) | 17 (17) | 10 (10)
Hemorrhage (Surgical and medical procedures) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT02952261/Prot_SAP_000.pdf